CLINICAL TRIAL: NCT01985321
Title: A Multicenter, Placebo-Controlled, Randomized, Double-Blind Study of the Safety and Efficacy of Merlin (Ethanol and Glycolic Acid Mixture) for the Episodic Treatment of Recurrent Herpes Labialis
Brief Title: Safety and Efficacy of Merlin (Ethanol and Glycolic Acid Mixture) for the Treatment of Cold Sores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topical Remedy (Industry)
Collaborators: Benu BioPharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR-H-211
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Recurrent Herpes Labialis
Keywords: herpes labialis; cold sore
MeSH Terms: conditions — Herpes Labialis | interventions — Ethanol; Neurofibromin 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Merlin - ethanol/glycolic acid solution (Experimental): 36 applications over a 96 hour period
  Interventions: Drug: ethanol/glycolic acid solution
- Placebo/Ethanol (Placebo Comparator): 36 applications over a 96 hour period
  Interventions: Drug: Placebo/Ethanol

INTERVENTIONS:
Drug: ethanol/glycolic acid solution — ethanol/glycolic acid solution
  Other Names: Merlin
  Arms: Merlin - ethanol/glycolic acid solution
Drug: Placebo/Ethanol — ethanol solution
  Other Names: Placebo
  Arms: Placebo/Ethanol

SUMMARY:
The purpose of this study is to determine if Merlin, a mixture of ethanol and glycolic acid, is safe and effective in the treatment of cold sores.

Subjects who meet the requirements to participate in the study will be put randomly, and equally, into one of two groups: 1) a group receiving Merlin to treat their cold sore; or 2)a group receiving a placebo of just ethanol to treat their cold sore. Neither the subject nor the site will know which treatment they will be getting. Once the subject has been assigned to a treatment group, they will be given a kit containing a bottle of the treatment and special swabs to apply the liquid. The subject will be told to take the kit home and wait until they think they are starting to get a cold sore.

Once a subject begins to feel something or see something that they think is the start of a cold sore, they are to immediately call the clinic. Once the clinic confirms that the subject is in fact starting to get a cold sore, the subject will be told to open the kit and begin treatment. From the start of treatment, there will be twelve (12) treatments, with either Merlin or placebo, applied six (6) hours apart, up to 3 per day, over the next 96 hours (4 days). Each treatment of Merlin or placebo is made up of three (3) applications given twenty (20) minutes apart, for a total of thirty-six (36) applications. FOr each application, the subject will use the special swab to put the Merlin or placebo solution on their cold sore.

Subjects will need to report daily to the clinic for a minimum of 3 consecutive days, until either the cold sore is completely healed or 14 days from the start of treatment, whichever comes first. At each clinic visit the cold sore will be observed to determine at what stage it is at or if it has healed. The subject will also be asked how they are feeling.

Subjects will also be told to record in a diary the time of each application of Merlin or placebo. They will also be asked to record how much pain, if any, related to the cold sore, that they are feeling.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18-75 years of age
* Female subjects must be using a medically acceptable form of birth control during the study. Acceptable birth control measures include, but are not limited to: abstinence, oral contraceptive pills or patch, injectable contraception, barrier contraceptives (condom, diaphragm with spermicide), IUD, vaginal contraceptive ring, surgical (hysterectomy, tubal ligation), vasectomized partner, and natural post-menopausal inability to conceive. Menopause is defined for this protocol as starting one year after the time of the last menstrual period.
* Subject must have a history of recurrent herpes labialis and report at least 3 separate recurrences (i.e. multiple herpetic lesions in one outbreak count as only one episode) during the preceding 12 months.
* Subject must have a history of experiencing prodromal symptoms of cold sores (e.g. itching, tingling, or burning) during at least half of their previous cold sore episodes.
* Subject must have a history of at least half of their cold sore episodes producing classical lesions (i.e., episodes that progressed through macule, papule, vesicle, crust, and healed).
* Subject must provide voluntary written informed consent to participate in this study.
* Subject is able to appear for a clinic visit within 24 hours from the time of treating cold sore and is able to return to the clinic for the full 14 day duration of the study if necessary.

Exclusion Criteria:

* Subjects with evidence of active malignancy or immunodeficiency disease within the last 30 days. Subjects who have completed therapy and are considered unlikely to relapse or who have had surgery and do not have any evidence of disease, are eligible for the study.
* Subject requires chronic use of immunomodifying drugs (e.g. systemic steroids) or topical steroids on or near the face; use of inhaled steroids does not exclude a subject from the study. If a subject is unlikely to get through the Treatment Phase of the protocol without requiring the use of an immunomodifying drug for a chronic condition the subject should be excluded.
* Subject requires chronic use of anti-viral medication.
* In females of childbearing potential, a positive urine pregnancy test at time of screening.
* Nursing mothers.
* Subject has abnormal skin conditions (e.g. acne, eczema, rosacea, psoriasis, albinism, or chronic vesiculobullous disorders) that occur in the area ordinarily affected by cold sores or has significant facial hair in the area of the cold sore that might affect the normal course of the cold sore or might impair accurate evaluation of the cold sore lesion.
* Subject has had a vaccine for herpes simplex virus type 1 (typically oral herpes) or 2 (typically genital herpes).
* Subject is currently enrolled in another clinical trial involving the use of a drug and/or a device.
* Subject requires chronic use of analgesics or non-steroidal anti-inflammatory agents (NSAIDs) except for low doses of aspirin (less than 325 mg/day) used for cardiovascular purposes. If a subject is unlikely to get through the Treatment Phase of the protocol without requiring the use of analgesia for a chronic condition, e.g. back pain, recurrent daily headaches, the subject should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Radiant Research, Santa Rosa, California
  - Radiant Research, Pinellas Park, Florida
  - Radiant Research, Chicago, Illinois
  - Radiant Research, Edina, Minnesota
  - Radiant Research, St Louis, Missouri
  - Radiant Research, Akron, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Radiant Reserach, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the start of the study in November of 2013 until the completion of the study in March 2014. There were 8 Investigators at 8 clinical sites.
Pre-assignment Details: There were no notable events or approaches for the study following enrollment, but prior to group assignment. Once subjects were found to meet the eligibility requirements at the screening/randomization visit they were randomized 1:1 into the active or placebo treatment groups.
Groups:
- Ethanol: 36 applications over a 96 hour period
Period: Overall Study
Arm/Group | Merlin - Ethanol/Glycolic Acid Solution | Ethanol
Started | 90 (This is Treatment Eligible Subjects only) | 83 (This is treatment eligible subjects only)
Completed | 79 | 78
Not Completed | 11 | 5
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 5 | 2
Not completed — Subject treated wrong type of sore | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population of the modified intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Merlin - Ethanol/Glycolic Acid Solution | Ethanol | Total
Number analyzed (Participants) | 89 | 83 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 74 | 147
  >=65 years | 16 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (15.54) | 48.6 (14.63) | 48.4 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 55 | 118
  Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 84 | 78 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 71 | 68 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 89 | 83 | 172

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessed Duration of Complete Healing of the Herpetic Episode
Time Frame: Days 1-14
Population: Modified Intent to Treat Population: 2 subjects in placebo group violated protocol and could not be evaluated for Complete Healing (83-2=81). 5 subjects in active group started treatment prior to contacting site; 1 subject in active group lost to follow-up with no site visits. These 6 active subjects not used in Complete Healing analysis (90-6=84)
Measure: Median (Full Range); unit: hours
Arm/Group | Merlin - Ethanol/Glycolic Acid Solution | Ethanol
Number analyzed (Participants) | 84 | 81
hours | 129.6 [38.9 to 334.2] | 154.6 [22.3 to 356.2]

2. Secondary Outcome: Number of Treatment Related Adverse Events
Time Frame: Days 1-28
Measure: Number; unit: participants
Arm/Group | Merlin - Ethanol/Glycolic Acid Solution | Ethanol
Number analyzed (Participants) | 89 | 83
participants | 9 | 3

ADVERSE EVENTS:
Time Frame: All subjects were followed daily until their cold sore lesion reached Stage 7, reporting daily for a minimum of 3 days, with the last clinic visit at the time of complete healing or at 14 days, whichever was earlier.
Arm/Group | Merlin - Ethanol/Glycolic Acid Solution | Ethanol
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/83
Other Adverse Events (participants affected / at risk) | 9/90 | 3/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merlin - Ethanol/Glycolic Acid Solution (N=90) | Ethanol (N=83)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 40 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and but can extend the embargo for up to 120 day to file patents or take other measures to preserve or secure its Intellectual Property.